CLINICAL TRIAL: NCT02467244
Title: Effect of Levothyroxine on Serum Adiponectin, Insulin Resistance and Cardiovascular Risk in Patients With Hypothyroidism
Status: Completed | Type: Observational
Sponsor: All India Institute of Medical Sciences, Bhubaneswar (Other)
Responsible Party: Principal Investigator, RITUPARNA MAITI, Associate Professor, All India Institute of Medical Sciences, Bhubaneswar
Other Study IDs: T/EM-F/Pharm/14/03
Record Dates: First submitted 2015-06-04; First posted 2015-06-10 (Estimated); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Hypothyroidism
Keywords: Hypothyroidism; Serum adiponectin; hsCRP; Homeostatic Model Assessment (HOMA-IR); Quantitative Insulin Sensitivity Check Index (QUICKI); Cardiovascular risk assessment scoring (Framingham scoring); Levothyroxin
MeSH Terms: conditions — Hypothyroidism | interventions — Thyroxine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Euthyroid group: Fifty (50) age and sex matched euthyroid subjects will serve as the control group. Control euthyroid subjects will be evaluated once at baseline and after 12 weeks.
- Hypothyroid group: Fifty (50) hypothyroid patients attending the outpatient department of General Medicine, AIIMS, Bhubaneswar, will be recruited for the present study following inclusion and exclusion criteria.
  Interventions: Drug: Levothyroxine

INTERVENTIONS:
Drug: Levothyroxine — At first visit, after taking detailed history including baseline symptomatology, clinical evaluation, and laboratory investigation, treatment will be started with levothyroxine (50 microgram/day). The dosage of levothyroxine (LT4) will be adjusted (at 4th and 8th week) in an attempt to keep the serum FT4 and TSH concentrations within the normal range. After 12 weeks, all the patients will be followed up, clinical and laboratory tests will be repeated.
  Groups: Hypothyroid group

SUMMARY:
The aim of this study is to evaluate plasma adiponectin level, insulin resistance, cardiovascular risk and their correlation (if any) in patients with hypothyroidism and also to investigate the effect of levothyroxine on these parameters. The study may explore the lacunae in present treatment protocol and can suggest the possibilities of add-on therapies for a better management.

DETAILED DESCRIPTION:
Hypothyroidism is associated with premature atherosclerosis and increased prevalence of coronary artery diseases. Long-term hypothyroidism is associated with severe cardiovascular manifestations including reduced intravascular volume, increased systemic vascular resistance, and hypertension. Hypothyroidism is one of the main causes of secondary dyslipidemia. The classic manifestations of hypothyroidism are raised VLDL, LDL and apo A. The increase in cardiovascular risk is not only due to dyslipidemia, but also to hemodynamic changes, endothelial dysfunction, hormonal and metabolic changes. Insulin resistance and the metabolic syndrome are important cardiovascular risk factors as insulin-resistant individuals with raised TSH have higher LDL concentrations.

Among the various markers associated with obesity and insulin resistance, of particular importance is adiponectin which is inversely related to the degree of adiposity, increases insulin sensitivity, and has antiatherogenic and anti-inflammatory properties, hence may be cardioprotective. Hypoadiponectinaemia is associated with obesity, insulin resistance and type II diabetes, as well as atherosclerosis, hypertension and coronary artery disease.

Treating hypothyroidism with levothyroxine has an antioxidant and cholesterol reducing effect, and thus already has proven beneficial impact on cardiovascular function, blood pressure and lipid profile. But the association of adiponectin and insulin resistance in hypothyroid state and future cardiovascular risk is still not clear because there are few published studies in this domain and result of some the studies are contradictory. The aim of this study is to evaluate plasma adiponectin level, insulin resistance, cardiovascular risk and their correlation (if any) in patients with hypothyroidism and also to investigate the effect of levothyroxine on these parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either sex, aged 18 years or above suffering from hypothyroidism (hypothyroidism was defined as serum TSH level > 5μIU/ml, serum FT3 level < 1.57 pg/ml, serum FT4 level < 0.7 ng/dL. Subclinical hypothyroidism was defined as an elevated TSH level and a normal serum FT3 and FT4 level) and need treatment (treatment is indicated in patients with TSH levels >10 µIU/mL or in patients with TSH levels between 5 and 10 µIU/mL in conjunction with goiter or positive anti-thyroid peroxidase antibodies (or both).
* Patients not having hepatic/renal dysfunction, Diabetes mellitus, and chronic inflammatory diseases and not taking any medications for thyroid disease.
* Euthyroid subjects not having any significant medical disease.

Exclusion Criteria:

* Patients with other comorbidites which can interfere the outcome measures.
* Patients who are already on levothyroxine therapy or taking other medications.
* Patients with subacute thyroiditis were excluded from the study since acute inflammation could influence the measurements.
* Pregnant and lactating mothers.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will be conducted on 50 patients of hypothyroidism attending the outpatient department of General Medicine, All India Institute of Medical Sciences, Bhubaneswar. Another 50 euthyroid, age-, sex-matched subjects will be recruited as control.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Change of Serum Adiponectin from baseline | At baseline and after 12 weeks at follow up
  Method: ELISA
Change of hsCRP from baseline | At baseline and after 12 weeks at follow up
  Method: ELISA
Change in Insulin resistance from baseline by Homeostatic Model Assessment (HOMA-IR) | At baseline and after 12 weeks at follow up

SECONDARY OUTCOMES:
Serum Insulin | At baseline and after 12 weeks at follow up
  Method: ELISA
Lipid profile (Total cholesterol) | At baseline and after 12 weeks at follow up
Lipid profile (LDL-C) | At baseline and after 12 weeks at follow up
Lipid profile (HDL-C) | At baseline and after 12 weeks at follow up
Lipid profile (Triglyceride) | At baseline and after 12 weeks at follow up
Long term glycemic status by Glycosylated hemoglobin (HbA1c%) | At baseline and after 12 weeks at follow up
Change in Insulin resistance from baseline by Quantitative Insulin Sensitivity Check Index (QUICKI) | At baseline and after 12 weeks at follow up
Change in Cardiovascular risk assessment scoring (Framingham scoring) from baseline | At baseline and after 12 weeks at follow up

CONTACTS AND LOCATIONS:
Overall Officials: DEBASISH HOTA, MD, DM, Study Director — AIIMS, Bhubaneswar
Locations (1):
- AIIMS, Bhubaneswar, Bhubaneshwar, Odisha, India

REFERENCES:
- [Result] Klein I, Ojamaa K. Thyroid hormone and the cardiovascular system. N Engl J Med. 2001 Feb 15;344(7):501-9. doi: 10.1056/NEJM200102153440707. No abstract available. PMID 11172193
- [Result] Benvenga S, Robbins J. Lipoprotein-thyroid hormone interactions. Trends Endocrinol Metab. 1993 Aug;4(6):194-8. doi: 10.1016/1043-2760(93)90116-v. PMID 18407156
- [Result] Fazio S, Palmieri EA, Lombardi G, Biondi B. Effects of thyroid hormone on the cardiovascular system. Recent Prog Horm Res. 2004;59:31-50. doi: 10.1210/rp.59.1.31. PMID 14749496
- [Result] Robinson K, Prins J, Venkatesh B. Clinical review: adiponectin biology and its role in inflammation and critical illness. Crit Care. 2011 Apr 20;15(2):221. doi: 10.1186/cc10021. PMID 21586104
- [Result] Maury E, Brichard SM. Adipokine dysregulation, adipose tissue inflammation and metabolic syndrome. Mol Cell Endocrinol. 2010 Jan 15;314(1):1-16. doi: 10.1016/j.mce.2009.07.031. Epub 2009 Aug 12. PMID 19682539
- [Result] Altinova AE, Toruner FB, Akturk M, Bukan N, Cakir N, Ayvaz G, Arslan M. Adiponectin levels and cardiovascular risk factors in hypothyroidism and hyperthyroidism. Clin Endocrinol (Oxf). 2006 Oct;65(4):530-5. doi: 10.1111/j.1365-2265.2006.02628.x. PMID 16984248
- [Result] Kowalska I, Borawski J, Nikolajuk A, Budlewski T, Otziomek E, Gorska M, Straczkowski M. Insulin sensitivity, plasma adiponectin and sICAM-1 concentrations in patients with subclinical hypothyroidism: response to levothyroxine therapy. Endocrine. 2011 Aug;40(1):95-101. doi: 10.1007/s12020-011-9446-5. Epub 2011 Mar 18. PMID 21424182